CLINICAL TRIAL: NCT06023992
Title: Compliance to Treatment in Adolescent Girls With Idiopathic Scoliosis: is it Associated With Perception of Appearance, Self-esteem, and Quality of Life?
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, İrem Çetinkaya, Lecturer, Halic University
Other Study IDs: karanki3
Record Dates: First submitted 2023-08-22; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent Idiopathic Scoliosis; perception of appearance; self-esteem; quality of life; compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Idiopathic scoliosis is a spinal deformity that occurs in adolescent girls and boys and is more progressive in girls. The cosmetic changes caused by the scoliotic spine cause negativity in perception of appearance and psychosocial problems in pubertal individuals, especially in girls. It is thought that brace used in conservative treatment increase this negativity in body image and affect compliance with treatment. In this study, it was aimed to determine whether there is an effect on the individual's compliance with the programmed treatment by investigating the perception of body appearance, self-esteem and quality of life of adolescent girls with idiopathic scoliosis. In this context, forty adolescent girls diagnosed with "idiopathic scoliosis" and followed in the "Formed Healthcare Scoliosis Unit" were included in the study. In the study, Walter Reed Visual Evaluation Scale was used to evaluate perception of appearance, Coopersmith Self-Esteem Inventory to evaluate self-esteem, and SRS-22 Scoliosis Patient Questionnaire to evaluate quality of life. Scoliosis Treatment Compliance Scale, which was developed by us and whose validity and reliability study was planned, was used to evaluate compliance with the treatment program.

DETAILED DESCRIPTION:
Scoliosis is a three-dimensional deformity of the spine in which a lateral deviation of more than 10º is observed in the coronal plane. Causes deterioration in sagittal, frontal and transverse planes; In scoliosis with lateral flexion, rotation and shortness components, there is a complex curvature of the spine.

The risk of progression, the initial degree of curvature, the age and maturation level of the patient are important for the treatment plan of a patient with AIS. In addition, cosmetic appearance and social factors play a role in the treatment protocol. Methods used in the treatment of scoliosis by considering the progression factor; observation, physiotherapy and specific rehabilitation, brace and surgical treatment.

There are studies showing that the results are positively affected if the programmed and recommended conservative treatment methods are complied with, and the importance of compliance to treatment is emphasized.

In order for the spinal tissues to respond to the forces created by the trunk orthoses (braces) used in the conservative treatment of AIS, a sufficient time and regular use of the brace is required. Studies have shown that there is non-compliance in the treatment process and that patients do not comply with the treatment, especially by not using their braces for a sufficient time during the day.

Exercise therapy has been used for years during follow-up and as a form of conservative therapy. Posture exercises (stabilization exercises) to provide spinal control, exercises to increase spinal flexibility (stretching exercises), exercises to correct muscle strength imbalance and to regulate breathing are applied. It has been reported that compliance with exercise therapy positively affects the treatment results.

It is very important to keep the treatment programs at home, to raise the awareness of the person to control the spine in daily life, to integrate the applied exercises into daily life activities and to support the scoliosis with sports activities. It is reported that correctly planned daily life activities and positions and sports activities that do not involve the risk of injury affect the treatment results positively.

The long treatment period in scoliosis, especially the use of braces, negatively affects daily life and increases the stress level. In this process, individuals with AIS may experience social isolation, depression, low participation in activities and non-compliance. It is mentioned that in order to achieve real success in treatment, the patient should come to terms with the situation he is in cognitively and psychosocial problems should be taken into account.

With the deviations in the frontal, sagittal and transverse planes of the scoliotic spine, the cosmetic effect becomes evident and negatively affects body image perception and psychological health. General physical changes in adolescence are accompanied by a reassessment of the young individual's self-concept. Studies have shown that compliance to treatment in individuals with AIS is associated with body image perceptions and self-esteem.

In addition, scoliosis is an important risk factor for poor quality of life in children and adolescents. It has been reported that the quality of life in AIS is significantly affected by the negative perception of the individual on body image, and low quality of life is associated with low self-esteem, especially in adolescent individuals who use braces.

When the literature is examined, studies examining the psychosocial effects of individuals with AIS and their relationships with quality of life and compliance to treatment are very limited. When the literature is examined, studies examining the psychosocial effects of individuals with AIS and their relationships with quality of life and compliance to treatment are very limited. When the measurement methods used in studies questioning adherence to treatment in the literature are examined, it is seen that there are limitations in the evaluation of corset and exercise therapy, as well as other treatment components such as daily life and sports activities. Since subjective and objective measurement methods are insufficient to question the treatment as a whole, a scale designed within the scope of this study was also presented to the literature. The aim of the investigators is to solve these limitations in the literature and to determine the effect of perception of deformity, self-esteem and quality of life on the adherence to treatment of the adolescent individual.

ELIGIBILITY:
Inclusion Criteria:

Provided that the family and the child volunteer to participate in the study,

* Being diagnosed with idiopathic scoliosis
* Girl gender,
* Be 12 years or older,
* Using and still wearing braces for at least 3 months due to AIS,
* Having been prescribed an exercise program

Exclusion Criteria:

* Having had previous spine surgery,
* Presence of a psychological or psychiatric diagnosis,
* Presence of any neurological, muscular, rheumatic or orthopedic diseases accompanying scoliosis.

Ages: 12 Years to 17 Years | Sex: Female
Age Groups: Child
Gender Based: Yes — In prevalence studies for AIS, it has been reported that the incidence in girls is higher than in boys. In addition, AIS is more progressive in girls and the need for treatment is greater than in boys.
Study Population: A clinic where individuals with scoliosis are treated and followed up by specialist physician and physiotherapists, as well as a scoliosis brace production and application center: Formed Healthcare Orthotics and Prosthesis Center - Scoliosis Unit.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2016-06-05 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Walter Reed Visual Assessment (WRVAS) | Baseline
  It is a valid scale consisting of 7 questions, each of which includes 5 visuals and evaluates the physical deformity perceived by the patients.The selected images are scored as the lowest "1" and the highest "5", and the highest total score is 35 and the lowest is 5. It is accepted that the higher the score, the more negative-evil perception of the deformity.
Coopersmith Self-Esteem Inventory | Baseline
  A valid and reliable short form of 25 questions adapted to children in the same age group was used to determine the level of self-esteem. Those who say 'No' to a negative statement and 'Yes' to a positive statement in the inventory get 1 point for each question. The level of self-esteem obtained is determined as "low" or "high" based on the average score of the group in which the person belongs.
Scoliosis Research Society-22 | Baseline
  It is a scoliosis-specific, valid and reliable quality of life scale that questions pain, body image perception, function/activity, mental health, and satisfaction with treatment. A minimum of 1 point (worst) and a maximum of 5 points (best) are taken for each question. Scoring is obtained by dividing the total score from each section by the number of questions in that section. As a result of the scoring, it is accepted that the higher the score, the higher the quality of life.
Scoliosis Treatment Compliance Scale | Baseline
  It is a scale prepared by us to evaluate compliance with the treatment program and recommended Activities of Daily Living in individuals with scoliosis. The patient can get a total of 28 points, with a minimum of 1 and a maximum of 4 points from each statement in the scale. It is observed that the higher the score, the higher the treatment compliance.

CONTACTS AND LOCATIONS:
Overall Officials: İrem Çetinkaya, MSc, Principal Investigator — Haliç University; Hürriyet G Yılmaz, MD, Study Chair — Haliç University; Melek G Yavuzer, MD, Study Director — Haliç University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pineda S, Bago J, Gilperez C, Climent JM. Validity of the Walter Reed Visual Assessment Scale to measure subjective perception of spine deformity in patients with idiopathic scoliosis. Scoliosis. 2006 Nov 8;1:18. doi: 10.1186/1748-7161-1-18. PMID 17090338
- [Result] Asher M, Min Lai S, Burton D, Manna B. Discrimination validity of the scoliosis research society-22 patient questionnaire: relationship to idiopathic scoliosis curve pattern and curve size. Spine (Phila Pa 1976). 2003 Jan 1;28(1):74-8. doi: 10.1097/00007632-200301010-00017. PMID 12544960
- [Result] Chan SL, Cheung KM, Luk KD, Wong KW, Wong MS. A correlation study between in-brace correction, compliance to spinal orthosis and health-related quality of life of patients with Adolescent Idiopathic Scoliosis. Scoliosis. 2014 Feb 22;9(1):1. doi: 10.1186/1748-7161-9-1. PMID 24559234
- [Result] Donzelli S, Zaina F, Negrini S. Compliance monitor for scoliosis braces in clinical practice. J Child Orthop. 2015 Dec;9(6):507-8. doi: 10.1007/s11832-015-0703-7. Epub 2015 Nov 2. No abstract available. PMID 26526180
- [Result] Helfenstein A, Lankes M, Ohlert K, Varoga D, Hahne HJ, Ulrich HW, Hassenpflug J. The objective determination of compliance in treatment of adolescent idiopathic scoliosis with spinal orthoses. Spine (Phila Pa 1976). 2006 Feb 1;31(3):339-44. doi: 10.1097/01.brs.0000197412.70050.0d. PMID 16449908
- [Result] Matamalas A, Bago J, D'Agata E, Pellise F. Body image in idiopathic scoliosis: a comparison study of psychometric properties between four patient-reported outcome instruments. Health Qual Life Outcomes. 2014 Jun 3;12:81. doi: 10.1186/1477-7525-12-81. PMID 24894714
- [Result] Meyer C, Haumont T, Gauchard GC, Leheup B, Lascombes P, Perrin PP. The practice of physical and sporting activity in teenagers with idiopathic scoliosis is related to the curve type. Scand J Med Sci Sports. 2008 Dec;18(6):751-5. doi: 10.1111/j.1600-0838.2007.00750.x. Epub 2008 Feb 2. PMID 18248544
- [Result] Negrini S, Antonini G, Carabalona R, Minozzi S. Physical exercises as a treatment for adolescent idiopathic scoliosis. A systematic review. Pediatr Rehabil. 2003 Jul-Dec;6(3-4):227-35. doi: 10.1080/13638490310001636781. PMID 14713590
- [Result] Negrini S, Aulisa AG, Aulisa L, Circo AB, de Mauroy JC, Durmala J, Grivas TB, Knott P, Kotwicki T, Maruyama T, Minozzi S, O'Brien JP, Papadopoulos D, Rigo M, Rivard CH, Romano M, Wynne JH, Villagrasa M, Weiss HR, Zaina F. 2011 SOSORT guidelines: Orthopaedic and Rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis. 2012 Jan 20;7(1):3. doi: 10.1186/1748-7161-7-3. PMID 22264320
- [Result] Rivett L, Stewart A, Potterton J. The effect of compliance to a Rigo System Cheneau brace and a specific exercise programme on idiopathic scoliosis curvature: a comparative study: SOSORT 2014 award winner. Scoliosis. 2014 May 30;9:5. doi: 10.1186/1748-7161-9-5. eCollection 2014. PMID 24926318
- [Result] Schwieger T, Campo S, Weinstein SL, Dolan LA, Ashida S, Steuber KR. Body Image and Quality-of-Life in Untreated Versus Brace-Treated Females With Adolescent Idiopathic Scoliosis. Spine (Phila Pa 1976). 2016 Feb;41(4):311-9. doi: 10.1097/BRS.0000000000001210. PMID 26555827